CLINICAL TRIAL: NCT06272032
Title: Prospective Multicenter Observational Study and Promotion of the Application of Focused Ultrasound in "Reduction of Hypertrophy" and "Desensitization" for Allergic Rhinitis
Brief Title: Prospective Multicenter Observational Study and Promotion of the Application of Focused Ultrasound in Allergic Rhinitis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yang Yucheng, Director, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023KFKT001
Record Dates: First submitted 2024-01-27; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; High-intensity focused ultrasound (HIFU); Clinical efficacy; safety
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Long-Term Synaptic Depression; Histamine Antagonists; Leukotriene Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity focused ultrasound (HIFU) (Active Comparator): The High-Intensity Focused Ultrasound (HIFU) knife, also known as the High-Intensity Focused Ultrasound Tumor Treatment System or HIFU ablation therapy, abbreviated as the HIFU knife, is a non-invasive and non-intrusive tumor treatment method utilizing "high-intensity focused ultrasound technology." This technology was successfully developed by the Ultrasound Medical Engineering Research Institute of Chongqing Medical University in 1997.
  Interventions: Procedure: High-intensity focused ultrasound (HIFU)
- Placebo (Placebo Comparator): For patients in the Placebo treatment group, treatment is provided based on the severity of their symptoms, following the protocols outlined in the Allergic Rhinitis (AR) diagnosis and treatment guidelines. Patients are administered intranasal corticosteroids, oral antihistamines, oral leukotriene receptor antagonists, and intranasal antihistamines, as appropriate, in accordance with the severity of their symptoms.
  Interventions: Drug: intranasal corticosteroids, oral antihistamines, oral leukotriene receptor antagonists, and intranasal antihistamines

INTERVENTIONS:
Procedure: High-intensity focused ultrasound (HIFU) — Ultrasound is a type of mechanical vibrational wave capable of penetrating living tissues without causing harm to the tissue. As a non-invasive physical modality, ultrasound boasts advantages such as non-invasive safety, excellent directional propagation, strong penetration capability, and optimal focusing effects. It can induce a series of structural and functional changes in tissue cells through actions like cavitation, mechanical force vibration, and heat generation, leading to corresponding clinical effects. Clinical studies have demonstrated that focused ultrasound not only improves symptoms of allergic rhinitis (AR) but also holds certain advantages in preserving the structural and functional integrity of the nasal mucosa.
  Other Names: Chongqing Haifu Technology Co., Ltd.
  Arms: High-intensity focused ultrasound (HIFU)
Drug: intranasal corticosteroids, oral antihistamines, oral leukotriene receptor antagonists, and intranasal antihistamines — intranasal corticosteroids, oral antihistamines, oral leukotriene receptor antagonists, and intranasal antihistamines and other therapies.
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a common condition, with nearly 300 million affected individuals in China, significantly impacting the quality of life. Despite standardized drug treatments, approximately 20% of AR patients experience inadequate control and require surgical intervention. AR manifests as nasal itching, sneezing, clear nasal discharge, nasal congestion, primarily associated with inflammation-induced hypertrophy of nasal turbinates and a heightened neurogenic state of the nasal mucosa. Surgical treatment focuses on "reducing hypertrophy" of nasal turbinates and "desensitizing" neurogenic hyperreactivity.High-intensity focused ultrasound (HIFU), as a minimally invasive therapeutic modality in AR, is still in its early stages of application and requires further multicenter clinical studies and widespread adoption. This project collaborates with six established institutions proficient in ultrasound treatment for AR. It aims to conduct a prospective multicenter observational study and subsequent dissemination, emphasizing the application of "reduction of hypertrophy" and "desensitization" in AR.Through standardized case selection, subjective and objective measures such as subjective symptom scores, quality of life assessments, nasal reflex, and nasal resistance tests before and after treatment will be employed to evaluate the effectiveness and safety of HIFU in "reducing hypertrophy" and "desensitizing" aspects of AR. Simultaneously, building on our established Otolaryngology Head and Neck Surgery Alliance and Southwest Allergy Alliance, the research results will be promoted through lectures, hands-on guidance, training sessions, academic conferences, and other means to facilitate the application of HIFU in AR and benefit a larger population of AR patients.

DETAILED DESCRIPTION:
Ultrasound is a form of mechanical vibrational wave that can penetrate living tissues without causing harm to the tissue. As a non-invasive physical modality, ultrasound boasts advantages such as non-invasive safety, excellent directional propagation, strong penetration capability, and optimal focusing effects. Through actions such as cavitation, mechanical force vibration, and heat generation, ultrasound can induce a series of structural and functional changes in tissue cells, resulting in corresponding clinical effects.As early as 2006, research reported that ultrasound, when focused at specific depths beneath the nasal mucosa, creates scattered, punctate coagulation-type necrosis in the biological focus zone beneath the mucosa. This process involves the dissolution and disappearance of nuclei in some vascular smooth muscle cells, endothelial cell degeneration, partial thrombosis formation, vacuolar degeneration of neural cells, and partial or complete necrosis of glandular cells. The coagulation-type necrosis subsequently dissolves and is absorbed, while the structure of nasal mucosa cup cells, ciliated columnar epithelial cells, and basal cells remains normal, without damage to cilia and microvilli.Clinical studies indicate that focused ultrasound not only improves symptoms of allergic rhinitis (AR) but also holds certain advantages in preserving the structural and functional integrity of the nasal mucosa. However, challenges exist in the current application of focused ultrasound for AR, including weak evidence from clinical studies, insufficient long-term efficacy observations, and limited understanding of treatment complications. Moreover, consensus is lacking on indications, treatment intensity, duration, safety, and complications avoidance, demanding urgent resolution.In light of these challenges and guided by the principle of "minimizing harm to patients in treatment," this study, centered on the minimally invasive surgical treatment of "reduction of hypertrophy" and "desensitization" in AR, aims to collaborate with six established tertiary hospitals in China proficient in ultrasound treatment for AR. The study will conduct a prospective multicenter clinical research to observe the clinical efficacy and safety of ultrasound focus in AR, explore its application value in AR, and promote the safe and effective clinical use of focused ultrasound in AR. The ultimate goal is to enhance the overall therapeutic effectiveness of AR, benefiting a large population of AR patients.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory AR.
2. Patients exhibiting persistent mucosal hypersensitivity or high secretion state (rhinorrhea, sneezing, etc.).

Exclusion Criteria:

1. Patients with exacerbation of nasal symptoms, uncontrolled or acute exacerbation of asthma
2. Patients with bleeding tendency, coagulation disorders
3. Patients with poor overall condition, unable to tolerate procedures
4. Patients with severe cardiovascular diseases, immune system disorders, malignant tumors
5. Patients with psychological disorders or poor compliance, combined with primary immunological diseases (such as Sjögren's syndrome) or abnormal results of tear secretion tests, etc.
6. Patients under 18 years of age or over 70 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Nasal Symptom Score | 1 month, 3 months, 6 months, 1 year, and 2 years post-treatment
  In accordance with the recommendations from the European Academy of Allergy and Clinical Immunology (EAACI), the primary assessment indicators for allergic rhinitis include scoring for four nasal symptoms (itchy nose, sneezing, runny nose, nasal congestion) and two ocular symptoms (itchy/sensation of foreign body/redness of eyes, tearing). Evaluation is conducted using the "four-point scale" and a Visual Analogue Score (VAS) to assess the individual symptoms and/or the overall nasal and ocular symptoms before, during, and after treatment.
  0 points: Asymptomatic
  1. point: Mild symptoms (Signs/symptoms noticeable but barely bothersome; easily tolerated)
  2. points: Moderate symptoms (Bothersome symptoms/signs that are clearly noticeable but tolerable)
  3. points: Severe symptoms (Intolerable, causing interference with daily activities and/or sleep)
daily medication score | 1 month, 3 months, 6 months, 1 year, and 2 years post-treatment
  The recorded information includes the medication name, method of use, and dosage. Symptomatic medication scoring is based on the patient's symptomatic medication usage, assessing clinical effectiveness. The scoring method employs a "three-step" approach: one point is assigned for the use of nasal, ocular, oral, or topical antihistamines; two points for nasal corticosteroids (or combined with antihistamines); and three points for oral corticosteroids (or combined with nasal steroids/antihistamines).
  1. point: Oral and/or topical antihistamines (nasal or ocular)
  2. points: Nasal corticosteroids (or combination with antihistamines)
  3. points: Oral corticosteroids (or combination with nasal corticosteroids/antihistamines)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Yang, Doctoral, Study Chair — Chongqing Medical University
Locations (1):
- Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan for this research project is designed to promote transparency, collaboration, and further scientific inquiry. In accordance with open science principles, we are committed to sharing anonymized individual participant data with other researchers who seek to validate findings, conduct meta-analyses, or explore related research questions.

REFERENCES:
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Seidman MD, Gurgel RK, Lin SY, Schwartz SR, Baroody FM, Bonner JR, Dawson DE, Dykewicz MS, Hackell JM, Han JK, Ishman SL, Krouse HJ, Malekzadeh S, Mims JW, Omole FS, Reddy WD, Wallace DV, Walsh SA, Warren BE, Wilson MN, Nnacheta LC; Guideline Otolaryngology Development Group. AAO-HNSF. Clinical practice guideline: Allergic rhinitis. Otolaryngol Head Neck Surg. 2015 Feb;152(1 Suppl):S1-43. doi: 10.1177/0194599814561600. PMID 25644617
- [Background] Bousquet J, Anto JM, Bachert C, Baiardini I, Bosnic-Anticevich S, Walter Canonica G, Melen E, Palomares O, Scadding GK, Togias A, Toppila-Salmi S. Allergic rhinitis. Nat Rev Dis Primers. 2020 Dec 3;6(1):95. doi: 10.1038/s41572-020-00227-0. PMID 33273461
- [Background] Wang XD, Zheng M, Lou HF, Wang CS, Zhang Y, Bo MY, Ge SQ, Zhang N, Zhang L, Bachert C. An increased prevalence of self-reported allergic rhinitis in major Chinese cities from 2005 to 2011. Allergy. 2016 Aug;71(8):1170-80. doi: 10.1111/all.12874. Epub 2016 Apr 13. PMID 26948849
- [Background] Bousquet J, Schunemann HJ, Togias A, Bachert C, Erhola M, Hellings PW, Klimek L, Pfaar O, Wallace D, Ansotegui I, Agache I, Bedbrook A, Bergmann KC, Bewick M, Bonniaud P, Bosnic-Anticevich S, Bosse I, Bouchard J, Boulet LP, Brozek J, Brusselle G, Calderon MA, Canonica WG, Caraballo L, Cardona V, Casale T, Cecchi L, Chu DK, Costa EM, Cruz AA, Czarlewski W, D'Amato G, Devillier P, Dykewicz M, Ebisawa M, Fauquert JL, Fokkens WJ, Fonseca JA, Fontaine JF, Gemicioglu B, van Wijk RG, Haahtela T, Halken S, Ierodiakonou D, Iinuma T, Ivancevich JC, Jutel M, Kaidashev I, Khaitov M, Kalayci O, Kleine Tebbe J, Kowalski ML, Kuna P, Kvedariene V, La Grutta S, Larenas-Linnemann D, Lau S, Laune D, Le L, Lieberman P, Lodrup Carlsen KC, Lourenco O, Marien G, Carreiro-Martins P, Melen E, Menditto E, Neffen H, Mercier G, Mosgues R, Mullol J, Muraro A, Namazova L, Novellino E, O'Hehir R, Okamoto Y, Ohta K, Park HS, Panzner P, Passalacqua G, Pham-Thi N, Price D, Roberts G, Roche N, Rolland C, Rosario N, Ryan D, Samolinski B, Sanchez-Borges M, Scadding GK, Shamji MH, Sheikh A, Bom AT, Toppila-Salmi S, Tsiligianni I, Valentin-Rostan M, Valiulis A, Valovirta E, Ventura MT, Walker S, Waserman S, Yorgancioglu A, Zuberbier T; Allergic Rhinitis and Its Impact on Asthma Working Group. Next-generation Allergic Rhinitis and Its Impact on Asthma (ARIA) guidelines for allergic rhinitis based on Grading of Recommendations Assessment, Development and Evaluation (GRADE) and real-world evidence. J Allergy Clin Immunol. 2020 Jan;145(1):70-80.e3. doi: 10.1016/j.jaci.2019.06.049. Epub 2019 Oct 15. PMID 31627910
- [Background] Jutel M, Agache I, Bonini S, Burks AW, Calderon M, Canonica W, Cox L, Demoly P, Frew AJ, O'Hehir R, Kleine-Tebbe J, Muraro A, Lack G, Larenas D, Levin M, Martin BL, Nelson H, Pawankar R, Pfaar O, van Ree R, Sampson H, Sublett JL, Sugita K, Du Toit G, Werfel T, Gerth van Wijk R, Zhang L, Akdis M, Akdis CA. International Consensus on Allergen Immunotherapy II: Mechanisms, standardization, and pharmacoeconomics. J Allergy Clin Immunol. 2016 Feb;137(2):358-68. doi: 10.1016/j.jaci.2015.12.1300. PMID 26853128
- [Background] Greiner AN, Hellings PW, Rotiroti G, Scadding GK. Allergic rhinitis. Lancet. 2011 Dec 17;378(9809):2112-22. doi: 10.1016/S0140-6736(11)60130-X. Epub 2011 Jul 23. PMID 21783242
- [Background] Cheng L, Chen J, Fu Q, He S, Li H, Liu Z, Tan G, Tao Z, Wang D, Wen W, Xu R, Xu Y, Yang Q, Zhang C, Zhang G, Zhang R, Zhang Y, Zhou B, Zhu D, Chen L, Cui X, Deng Y, Guo Z, Huang Z, Huang Z, Li H, Li J, Li W, Li Y, Xi L, Lou H, Lu M, Ouyang Y, Shi W, Tao X, Tian H, Wang C, Wang M, Wang N, Wang X, Xie H, Yu S, Zhao R, Zheng M, Zhou H, Zhu L, Zhang L. Chinese Society of Allergy Guidelines for Diagnosis and Treatment of Allergic Rhinitis. Allergy Asthma Immunol Res. 2018 Jul;10(4):300-353. doi: 10.4168/aair.2018.10.4.300. PMID 29949830
- [Background] Zhong B, Li LK, Deng D, Du JT, Liu YF, Liu F, Liu SX. Effect of High-Intensity Focused Ultrasound Versus Plasma Radiofrequency Ablation on Recurrent Allergic Rhinitis. Med Sci Monit. 2019 Sep 9;25:6775-6781. doi: 10.12659/MSM.916228. PMID 31496537